CLINICAL TRIAL: NCT03709966
Title: Using a Portable Monitoring Device to Increase Motivation for Physical Activity in Patients with Type 2 Diabetes
Brief Title: Portable Monitoring Device, Physical Activity Motivation and Patients with Type 2 Diabetes
Acronym: DBFitbit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Caroline Rhéaume, Principal investigator, MD, PhD, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-2018-07
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2; Physical Activity; Motivation
Keywords: Portable monitoring device
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: The methodology used for this study consists of a pilot randomized controlled trial of 30 Type 2 diabetes patients already followed by health professionals from GMF-U Quatre-Bourgeois
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- FitBit (Experimental): Portable technological support to monitor physical activity, similar to a wrist-sport watch with many features including step calculations, distance traveled, calories burned, but also heart rate and sleep status.
  Interventions: Device: Portable monitoring device
- Routine (Active Comparator): Physical activity promotion supported by a kinesiologist
  Interventions: Behavioral: Routine

INTERVENTIONS:
Device: Portable monitoring device — similar to a wrist-sport watch with many features including step calculations, distance traveled, calories burned, but also heart rate and sleep status
  Other Names: FitBit
  Arms: FitBit
Behavioral: Routine — Physical activity promotion supported by a kinesiologist
  Other Names: PA promotion
  Arms: Routine

SUMMARY:
The intervention proposed for this project aims to improve the practice of physical activity (PA) for people with type 2 diabetes by increasing their motivation using a portable device to monitor PA (FitBit). This study will provide preliminary data to assess the feasibility of the intervention, its acceptability for patients with type 2 diabetes, and its potential impact of PA motivation and PA level.

DETAILED DESCRIPTION:
It is recognized that the adoption of healthy lifestyle habits, such as the practice of physical activity (PA) on a regular and constant basis, contributes significantly to reducing the prevalence of diabetes and its complications. The use of portable technological support to monitor PA can contribute to a favorable behavioral change in people with chronic diseases such as diabetes. Objective: The intervention proposed for this project aims to improve the practice of PA for people with type 2 diabetes, by increasing their motivation using a portable device tracking of PA (FitBit). The device is similar to a wrist-sport watch with many features including step calculations, distance traveled, calories burned, but also heart rate and sleep status. The information recorded by the watch can be synchronized and transmitted directly to the FitBit application, allowing it to be viewed and tracked on a daily basis, and also the ability to produce weekly and monthly reports and adjust personal goals. Methods: This study consists in a pilot randomized controlled trial of 30 Type 2 diabetes patients already followed by health professionals from a University-affiliated Family Medicine Group (GMF-U Quatre-Bourgeois). Patients are randomly assigned to one of these two conditions: routine follow-up, including a PA promotion intervention supported by a kinesiologist from the research center of the Institut de cardiologie et de pneumologie de Québec (CRIUCPQ) or FitBit follow-up, which consists of routine follow-up with the adding the portable PA tracking device. We plan to recruit 15 patients per group. The randomization is done by a statistician from CRIUCPQ. Inclusion and Exclusion Criteria: To participate in the study, participants must meet the following inclusion criteria: to be in a stable medical condition, sedentary and type 2 diabetic man or woman between the ages of 18 and 90 years of age. People with acute renal failure, FG below 30 ml and those under 18 years of age are excluded. Intervention: The intervention lasts 3 months and involves a total of 3 appointments. The first appointment takes place with the physician in charge of the study in order to evaluate the patient's record and to validate their eligibility. The glycated hemoglobin data and cardiometabolic measurements taken by the attending physician of each participant will be collected by the physician and clinical researcher in charge of the project. These same measures will be taken at the 3-month follow-up prescribed to each participant and this data will be collected a second and last time by the physician in charge of the project, at the very end of the intervention. Following their visit to the physician in charge of the study, the participants will meet the research professional who will be responsible for explaining the project in more details and obtaining their consent. The second appointment is attended by a kinesiologist who will distribute a physical activity motivation questionnaire, a physical activity questionnaire and a logbook to the participants. A personalized physical activity program will also be proposed to all participants. At the 6th week of the intervention, the kinesiologist will follow up with all participants to verify the integration of the physical activity program. A third appointment is planned at the very end of the intervention with the kinesiologist. Participants will be asked to complete the same questionnaires as for visit # 2 and submit their completed logbook. The participants in the experimental group will have a satisfaction questionnaire / appreciation of the technology to be completed in addition to the other questionnaires. They will also have to bring back their Fitbit material during this appointment.

ELIGIBILITY:
Inclusion Criteria:

* To be in a stable medical condition, sedentary, type 2 diabetic man or woman between the ages of 18 and 90 years of age

Exclusion Criteria:

* People with acute renal failure FG below 30 ml and those under 18 years of age.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Physical activity measurements | 3 months
  Godin Leisure-Time Exercise Questionnaire

SECONDARY OUTCOMES:
Motivation and auto-regulation of physical activity | 3 months
  Behavioral Regulation in Exercise Questionnaire (BREQ) version 2

OTHER OUTCOMES:
Acceptability, satisfaction of the portable monitoring device and compliance | 3 months
  Homade questionnaire with 10 questions
Cardiometabolic measurements: glycated hemoglobin | Before and after the clinical intervention: 3 months
  Blood test
Cardiometabolic measurements: systolic and diastolic blood pressure | Before and after the clinical intervention: 3 months
  Taken with standard apparel
Cardiometabolic measurements: Weight | Before and after the clinical intervention: 3 months
  measured with a bioimpedance balance InBody
Cardiometabolic measurements: fat percentage | Before and after the clinical intervention: 3 months
  measured with a bioimpedance balance InBody
Cardiometabolic measurement: Triglycerides | Before and after the clinical intervention: 3 months
  Blood test
Cardiometabolic measurement: High-density lipoprotein cholesterol (HDL) | Before and after the clinical intervention: 3 months
  Blood test
Cardiometabolic measurement: Low-density lipoprotein cholesterol (LDL) | Before and after the clinical intervention: 3 months
  Blood test

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Rhéaume, MD-PhD, Principal Investigator — Laval University; Caroline Rhéaume, MD-PhD, Study Director — Laval University
Locations (1):
- GMF-UMF Laval-Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pelletier C, Chabot C, Gagnon MP, Rheaume C. Implementing an Activity Tracker to Increase Motivation for Physical Activity in Patients With Diabetes in Primary Care: Strengths, Weaknesses, Opportunities and Threats (SWOT) Analysis. JMIR Form Res. 2023 Mar 10;7:e44254. doi: 10.2196/44254. PMID 36897642